CLINICAL TRIAL: NCT06718322
Title: Towards Large-Scale Adaptation and Tailored Implementation of Primary Cancer Prevention Programs Across 9 Countries
Brief Title: PIECES - Towards Large-Scale Adaptation and Tailored Implementation of Primary Cancer Prevention Programs
Acronym: PIECES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hidde van der Ploeg (Other)
Collaborators: Helse Bergen Hospital Trust (Unknown); Stichting Trimbos-Instituut (Other); Hannover Medical School (Other); Universiteti i Tiranes (Other); Public Health Center of MOH of Ukraine (Unknown); German Cancer Research Center (Other); University of Stirling (Other); University of Limerick (Other); The University of Queensland (Other); Institut Català d'Oncologia (Other); Istituto per lo Studio, la Prevenzione e la Rete Oncologica (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); Dreamedsoft Solutions (Unknown); German Network for Tobacco Free Healthcare Services (Unknown)
Responsible Party: Sponsor-Investigator, Hidde van der Ploeg, Professor, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Project 101104390
Record Dates: First submitted 2024-11-13; First posted 2024-12-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-10

CONDITIONS: Focus of Study: Tailored Implementation
Keywords: PIECES; Tailored implementation; Implementation support; PCP-IT; Primary Cancer Prevention

STUDY DESIGN:
Intervention Model Description: This study evaluates an implementation intervention targeting professionals implementing a cancer prevention program. The intervention is an online toolkit that supports implementers in selecting and adapting an evidence-based cancer prevention program and developing a tailored implementation plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Local implementation teams (Experimental): The local implementation teams for this study, referred to as the implementers of the Primary Cancer Prevention Implementation Toolkit (PCP-IT), are the primary users of the toolkit and play a central role in tailoring and implementing cancer prevention interventions. Each team is responsible for selecting and adapting the intervention to meet local needs and developing a tailored implementation plan. Each team is led by an implementation lead, who directly oversees the implementation process and ensures the team effectively uses the PCP-IT to guide their work. In some cases, the implementation lead may also serve as the implementation coordinator. The coordinator's role is to provide higher-level oversight and may involve coordinating multiple implementation teams across various locations, such as hospitals, or focusing on a single team at one site.
  Interventions: Other: Primary Cancer Prevention Implementation Toolkit (PCP-IT)

INTERVENTIONS:
Other: Primary Cancer Prevention Implementation Toolkit (PCP-IT) — The PCP-IT is an online implementation support toolkit which aims to support implementation teams in improving the implementation of primary cancer prevention programs (PCPs). The PCP-IT builds upon the theory-base and the proven to be effective ItFits tool. The PCP-IT encompasses a total of six modules which are designed to guide implementers through the process of selecting and adapting PCP programs, identifying and addressing barriers, and developing and applying tailored implementation strategies. The toolkit includes: (1) a repository of PCP programs, (2) a repository of determinants of practice, (3) a repository of implementation strategies, (4) stakeholder consultation at all stages, (5) an online community of implementation practitioners, and (6) structured stepped process flows, instructions, examples and worksheets for working with the materials. https://global.itfits-toolkit.com/

SUMMARY:
The PIECES project aims to evaluate the Primary Cancer Prevention Implementation Toolkit (PCP-IT), an online implementation support toolkit that aids implementation teams in improving the implementation of primary cancer prevention programs (PCPs).

The primary aim of the PIECES study is to support and learn from the process of selecting, adapting, and implementing existing evidence-based programs to improve implementation outcomes and by that, improve the reach and effectiveness of primary cancer prevention programmes in real-world settings.

The study objectives are:

1. To assess whether the PCP-IT is usable and if implementation teams are satisfied with the tool;
2. To assess what works for whom in using the PCP-IT for selecting, adapting, and implementing PCP programs;
3. To assess whether the PCP-IT is feasible and effective in improving acceptability, adoption, penetration, and sustainable implementation of the PCP programs.

The PCP-IT will be used by various implementation settings across 9 countries (8 European countries and Australia). A multi-site case comparison design is used to generate in-depth knowledge about the performance and working mechanisms of the PCP-IT. Similarities, differences, and patterns across the different implementation sites will be investigated using a Realist Evaluation approach.

DETAILED DESCRIPTION:
A range of modifiable factors are associated with cancer incidence among the population of the European Union (EU) and beyond. These include: 1) tobacco smoking and exposure to second-hand smoke, 2) alcohol consumption, 3) poor physical activity, 4) HPV infection, 5) sun exposure, and 6) poor diet. Various Primary Cancer Prevention (PCP) programs are currently available to address these risk factors with proven effectiveness. Decision-makers and implementers face the challenge of: 1) selecting appropriate and suitable programs, 2) tailoring the programs to the local context and consulting stakeholders, and 3) developing a tailored plan (i.e., strategies) for effectively implementing the selected and adapted PCP program. The lack of guidance and support for this complex and time-consuming process leads to two undesired outcomes: 1) the selection of ineffective or poorly adapted PCP programs, and 2) the application of ineffective implementation strategies that do not target local and context-dependent barriers to implementation. These scenarios are likely to reduce the effectiveness of primary cancer prevention programs in real-world settings, leading to inefficiencies and failing to prevent new cancer cases.

The PIECES project involves the development and evaluation of an online implementation support toolkit (the Primary Cancer Prevention Implementation Toolkit (PCP-IT)). The PCP-IT aims to support implementation teams in improving the implementation of primary cancer prevention programs (PCPs). The PCP-IT builds upon the theory-base and the proven to be effective ItFits tool. The PCP-IT encompasses a total of six modules. The modules are designed to guide implementers through the process of selecting and adapting PCP programs, identifying and addressing barriers, and developing and applying tailored implementation strategies. The core resources contributing to the generative mechanisms of the toolkit include: 1) a repository of primary cancer prevention programs, 2) a repository of determinants of practice, 3) a repository of implementation strategies, 4) stakeholder consultation at all stages, 5) an online community of implementation practitioners, and 6) structured stepped process flows, instructions, examples and worksheets for working with the materials.

In the PIECES study, a multi-site case comparison design is chosen to generate in-depth knowledge about the performance and working mechanisms of the PCP-IT. Similarities, differences, and patterns across the cases (i.e. different implementation settings) will be investigated using a Realist Evaluation approach. A pre/post-test measure will be applied to descriptively assess implementation outcomes. A time horizon of two years is selected to assess change over time.

The PCP-IT will be used in various countries and implementation settings, aiming for a rich representation of healthcare systems (Spain, the Netherlands, Albania, the United Kingdom, Ireland, Italy, Ukraine, Germany (3 settings), and Australia).

Within each implementation site, different types of participants with specific roles can be distinguished:

1. implementation coordinator: oversees the implementation process and can coordinate one or multiple implementation teams.
2. implementation lead: oversees the implementation process of one implementation team and is part of that team. This person is responsible for working through the PCP-IT with their implementation team. It is possible that the implementation coordinator and implementation lead is the same person.
3. implementation core team: the implementation team consists of the toolkit users who are the group responsible for selecting and adapting the PCP, as well as developing a tailored implementation plan.
4. service deliverers: the team/persons responsible for the actual implementation of the selected PCP and tailored implementation strategies.

The PCP-IT will be evaluated through various levels of evalution, with a primary focus on evaluating the use of the PCP-IT and implementation outcomes of the PCP programs.

1. PCP-IT: evaluating the use of the PCP-IT by the implementation teams.
2. PCP implementation: evaluating implementation outcomes of the implemented PCP programs
3. PCP impact: evaluating the impact of the implemented PCP programs (in terms of changes in behaviour the PCP program is targeting) (conducted if feasible).

The primary focus of the evaluation study will be on evaluating the use of the PCP-IT (level 1) and the implementation outcomes of the PCP program (level 2). Level 3 evaluation, which involves evaluating the impact of the implemented PCP programs on targeted behavior changes, is not part of the central evaluation study. However, implementation sites are encouraged to conduct level 3 evaluations if resources such as time and funding permit. While level 3 evaluation is not critically necessary from a research perspective-since PCP programs included in the PCP-IT repository have already demonstrated effectiveness-it is important from a monitoring perspective. Conducting level 3 evaluations can for example help implementation sites to:

* Assess whether the adapted PCP programs are achieving the desired outcomes
* Provide ongoing feedback to refine and improve the programs, ensuring the programs remain effective and relevant
* Show stakeholders, including funders and participants, that the programs are making a tangible difference, thereby justifying continued support and investment.

For this third level of evaluation, the specific details and ethical approvals are managed by each local implementation site. However, recommendations grounded in previous research are provided to guide the process and help maintain consistency across sites.

ELIGIBILITY:
Inclusion Criteria:

* User of the PCP-IT, involved in implementation of PCP programs.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Competencies in Implementation | Month 0, repeated every six months until month 24.
  Participants are asked to rate how skilled they feel in various implementation competencies. Respondents evaluate their skills for each item on a 5-point Likert scale, ranging from not at all to extremely (not at all, slightly, moderately, very, extremely).

SECONDARY OUTCOMES:
Organizational Readiness for Implementing Change (ORIC) | Month 0, repeated every six months until month 24.
  Participants are asked to indicate how they perceive the readiness of their organization to implement a cancer prevention program. This is assessed using the Organizational Readiness for Implementing Change (ORIC) instrument, which includes 12 items about an organizational readiness to implement a cancer prevention program. Respondents rate their level of agreement with each item on a 5-point Likert scale, ranging from I disagree to I agree (I disagree, I somewhat, disagree, Neither agree nor disagree, I somewhat agree, I agree).
Perceived Ease of Use | Month 6, repeated every six months until month 24.
  Participants are asked to indicate their agreement with 4 items about how useful they perceive the toolkit to be in their job. This is assessed using the Perceived Ease of Use instrument. Respondents rate their level of agreement with each item on a 7-point Likert scale, ranging from I strongly disagree to I strongly agree (I strongly disagree, I disagree I somewhat, disagree, Neither agree nor disagree, I somewhat agree, I agree, I strongly agree).
Perceived Usefulness | Month 6, repeated every six months until month 24.
  Participants are asked to indicate their agreement with 4 items about how easy they think it is to work with the toolkit. This is assessed using the Perceived Usefulness instrument. Respondents rate their level of agreement with each item on a 7-point Likert scale, ranging from I strongly disagree to I strongly agree (I strongly disagree, I disagree I somewhat, disagree, Neither agree nor disagree, I somewhat agree, I agree, I strongly agree).
Satisfaction with the PCP-IT | Month 6, repeated every six months until month 24.
  Participants are asked to rate their satisfaction with the toolkit using a Visual Analogue Scale (VAS). Respondents provide a score reflecting their satisfaction with specific modules or components of the toolkit. The VAS ranges from 0 to 10, where 0 represents no satisfaction, 5 represents neutral, and 10 represents extreme satisfaction.
Perceived impact of the PCP-IT | Month 6, repeated every six months until month 24.
  Participants are asked to rate the extent to which they think the toolkit has contributed to various implementation steps using a Visual Analogue Scale (VAS). The VAS ranges from 0 to 10, where 0 represents non-existent, 5 represents somewhat, and 10 represents very much.
Behavioral Intention | Month 6, repeated every six months until month 24.
  Participants are asked to indicate their agreement with 4 items about their intention or likelihood of using the toolkit in the future. This is assessed using the Behavioral Intention instrument. Respondents rate their level of agreement with each item on a 7-point Likert scale, ranging from I strongly disagree to I strongly agree (I strongly disagree, I disagree I somewhat, disagree, Neither agree nor disagree, I somewhat agree, I agree, I strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Femke van Nassau, PhD, Study Chair — Amsterdam UMC
Locations (11):
- Universiteti i Mjekesise Tirane, Tirana, Albania
- The University of Queensland, Saint Lucia, Australia
- Germany (3):
  - German Network for Tobacco Free Healthcare Services, Berlin
  - Hannover Medical School, Hanover
  - German Cancer Research Center (DFKZ), Heidelberg
- University of Limerick, Limerick, Ireland
- ISPRO, Florence, Italy
- Trimbos Instituut, Utrecht, Netherlands
- Catalan Institute of Oncology, Barcelona, Spain
- State Institution Public Health Center of the Ministry of Health of Ukraine, Kyiv, Ukraine
- University of Stirling, Stirling, United Kingdom

REFERENCES:
- [Background] Vis C, Schuurmans J, Aouizerate B, Atipei Craggs M, Batterham P, Buhrmann L, Calear A, Cerga Pashoja A, Christensen H, Dozeman E, Duedal Pedersen C, Ebert DD, Etzelmueller A, Fanaj N, Finch TL, Hanssen D, Hegerl U, Hoogendoorn A, Mathiasen K, May C, Meksi A, Mustafa S, O'Dea B, Oehler C, Piera-Jimenez J, Potthoff S, Qirjako G, Rapley T, Rosmalen J, Sacco Y, Samalin L, Skjoth MM, Tarp K, Titzler I, Van der Eycken E, van Genugten CR, Whitton A, Zanalda E, Smit JH, Riper H. Effectiveness of Self-guided Tailored Implementation Strategies in Integrating and Embedding Internet-Based Cognitive Behavioral Therapy in Routine Mental Health Care: Results of a Multicenter Stepped-Wedge Cluster Randomized Trial. J Med Internet Res. 2023 Feb 3;25:e41532. doi: 10.2196/41532. PMID 36735287
- [Background] Padek M, Colditz G, Dobbins M, Koscielniak N, Proctor EK, Sales AE, Brownson RC. Developing educational competencies for dissemination and implementation research training programs: an exploratory analysis using card sorts. Implement Sci. 2015 Aug 12;10:114. doi: 10.1186/s13012-015-0304-3. PMID 26264453
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- See also: Project Website — https://pieces-project.eu/